CLINICAL TRIAL: NCT01017757
Title: Cross-sectional Analysis of Subclinical Interstitial Lung Abnormalities in Stable Renal Transplant Recipients by High-resolution CT Scan
Brief Title: Interstitial Lung Abnormalities in Renal Transplant Recipients
Acronym: LCRT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Parma (Other)
Responsible Party: Carlo Buzio, University of Parma
Other Study IDs: LungCtRenalTx
Record Dates: First submitted 2009-11-18; First posted 2009-11-23 (Estimated); Last update posted 2009-11-23 (Estimated); Status verified 2009-11

CONDITIONS: Renal Transplantation; Kidney-pancreas Transplantation
Keywords: Interstitial lung disease; Immunosuppressive therapy; Renal transplant
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Renal transplant patients
  Interventions: Procedure: High-resolution CT scanning

INTERVENTIONS:
Procedure: High-resolution CT scanning — High-resolution CT scanning

SUMMARY:
Immunosuppressive drugs such as tacrolimus, cyclosporine, mycophenolate mofetil, sirolimus and everolimus may have toxic pulmonary effects, particularly interstitial alterations. The aim of the present study is to explore the presence of subclinical interstitial lung abnormalities in stable renal transplant recipients taking the different immunosuppressive drugs used as maintenance therapy for renal transplantation.

DETAILED DESCRIPTION:
Prospective, cross-sectional study examining the high-resolution CT scans obtained in 63 stable renal transplant recipients taking immunosuppressive treatment for at least 24 months. The findings in patients taking the newer immunosuppressive drugs (mycophenolic acid, sirolimus and everolimus) are compared with those of the patients treated in the traditional way (cyclosporine, tacrolimus, azathioprine). All patients undergo high-resolution CT scanning.

Eligibility criteria: recipients of kidney or kidney-pancreas transplant, on immunosuppressive therapy for at least 24 months, with stable renal function and absence of any overt lung disease or lung alterations induced by other drugs, systemic diseases or occupational exposure to fibrogenic agents.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant patients with stable renal function taking immunosuppressive therapy for at least 24 months and providing written informed consent to participate to the study

Exclusion Criteria:

* Overt lung disorders, lung toxicity due to other drugs or occupational exposure to lung-toxic agents
* Systemic connective tissue disorders or systemic vasculitis

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney or kidney-pancreas recipients, on immunosuppressive therapy for at least 24 months
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2007-06; Primary Completion 2007-10 (Actual); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Subclinical lung alterations as assessed by high-resolution CT scanning | CT is performed at study entry and, if abnormalities are found, it is repeated at 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Buzio, MD, Principal Investigator — University of Parma
Locations (1):
- Department of Clinical Medicine Nephrology and Health Science, Parma University Hospital, Parma, Parma, Italy